CLINICAL TRIAL: NCT03061903
Title: Closed Incision Negative Pressure Therapy vs. Standard of Care for Surgical Incision Management in High-Risk Patients Following Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Closed Incision Negative Pressure Therapy vs Standard of Care
Acronym: Prevena
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Principal Investigator, Roshan P. Shah, Assistant Professor of Orthopedic Surgery at the Columbia Univer, Dept of Orthopaedic Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR5849
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Wound Complication
Keywords: total hip arthroplasty; direct anterior approach; wound complication

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either the ciNPT intervention group (Prevena) or the control group (Aquacel) using computer-generated, randomized envelopes with equal numbers in each treatment arm. Both dressings will be applied under sterile conditions at the end of the THA surgery, while still in the operating room, and then removed after 7 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prevena (Experimental): Subjects will receive PREVENA after surgery.
  Interventions: Device: Prevena
- Aquacel (Active Comparator): Subjects will receive AQUACEL Ag after surgery.
  Interventions: Device: Aquacel

INTERVENTIONS:
Device: Prevena — Closed Incision Negative Pressure Therapy (bandage over the incision sealed with negative pressure of a vacuum) to be placed on after surgery for 7 days.
  Prevena™, by KCI, is currently being used selectively in high-risk patients and a FDA-approved device.
  Other Names: Closed incision negative pressure therapy; ciNPT
  Arms: Prevena
Device: Aquacel — Water resistant, silver-impregnated, antimicrobial hydrofiber dressing that is placed on after surgery for 7 days.
  AQUACEL® Ag, by Convatec, is currently the standard of care for postoperative wound dressing and a FDA-approved device.
  Other Names: Aquacel Ag
  Arms: Aquacel

SUMMARY:
High risk patients who receive direct anterior approach total hip arthroplasty are more likely to experience wound complications. The purpose of this study is to determine whether the usage of closed incision negative pressure dressings decreases the risk of wound complication compared to standard dressings. Patients who decide to participate in the study will be randomized to one of the two dressing prior to surgery and will leave the operating room with one of the treating dressings. Patient will be monitored 90 days after surgery for wound complications and pictures of the wounds will be taken. The patients course of treatment besides being randomized to one of the two dressings will be identical to any other patient received a Direct Anterior Approach for Total Hip Arthroplasty (DAA THA).

The primary outcome measure will be uneventful wound healing (requiring no intervention) versus the occurrence of wound complications (wound drainage, breakdown, necrosis, dehiscence, superficial or deep infection) requiring additional intervention. Intervention will be defined as any attempt of the surgeon to improve wound healing (in-office debridement, topical ointment, aspiration, antibiotic therapy, or return to the OR for the wound). Secondary outcome measures will include duration of wound healing delay, length of hospital stay, number of days of antibiotic therapy, and direct and estimated indirect costs.

DETAILED DESCRIPTION:
The goal of this study is to determine the efficacy of closed incision negative pressure therapy (CiNPT) for prevention of wound complications and return to the operating room for wound complications in patients with pre-determined risk factors that affect wound healing. This is will be a prospective, randomized, controlled trial. Subjects will be randomly assigned to either the ciNPT intervention group or the control group using computer-generated, randomized envelopes with equal numbers in each treatment arm. Both dressings will be applied under sterile conditions at the end of the DAA THA surgery, while still in the operating room, and then removed after 7 days.

Patients randomized to the control group will receive a conformable, water resistant, silver-impregnated, antimicrobial hydrofiber dressing (AQUACEL® Ag, Convatec) which is currently the standard of care at our institution for postoperative wound dressing. This dressing is left in place for 7 days and then removed by the patient or visiting nurse at home. Patients randomized to the study group will receive an incisional ciNPT device, which is currently being used selectively in high-risk patients at our institution (Prevena™, KCI). Both wound dressings are FDA-approved devices. Due to the obvious difference in appearance of the two dressings, neither patients nor treating surgeons can be blinded to treatment arm.

Wounds will be assessed postoperatively at regular intervals until wound healing is achieved. This will occur at least 2 and 6 weeks after surgery, which are standard intervals in our current postoperative protocol. No additional office visits will be needed for patients in the control or treatment arms. Photodocumentation of the wounds will occur at two and six weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing primary total hip arthroplasty (THA) through a direct anterior approach by one of the investigating surgeons; and
2. The presence of one or more of these risk factors for delayed or problematic wound healing:

   1. Diabetes
   2. Obesity (Body Mass Index (BMI) > 30)
   3. Active smoking
   4. Previous Hip Surgery

Exclusion Criteria:

1. Patients undergoing primary THA through a different approach
2. Patients undergoing primary THA through a direct anterior approach but without any of the above risk factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshan P Shah, MD, Principal Investigator — Columbia University
Locations (3):
- United States (2):
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
- Humber River Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jewett BA, Collis DK. High complication rate with anterior total hip arthroplasties on a fracture table. Clin Orthop Relat Res. 2011 Feb;469(2):503-7. doi: 10.1007/s11999-010-1568-1. PMID 20886324
- [Background] Christensen CP, Karthikeyan T, Jacobs CA. Greater prevalence of wound complications requiring reoperation with direct anterior approach total hip arthroplasty. J Arthroplasty. 2014 Sep;29(9):1839-41. doi: 10.1016/j.arth.2014.04.036. Epub 2014 May 2. PMID 24890998
- [Background] Jahng KH, Bas MA, Rodriguez JA, Cooper HJ. Risk Factors for Wound Complications After Direct Anterior Approach Hip Arthroplasty. J Arthroplasty. 2016 Nov;31(11):2583-2587. doi: 10.1016/j.arth.2016.04.030. Epub 2016 May 6. PMID 27267230
- [Background] Pulido L, Ghanem E, Joshi A, Purtill JJ, Parvizi J. Periprosthetic joint infection: the incidence, timing, and predisposing factors. Clin Orthop Relat Res. 2008 Jul;466(7):1710-5. doi: 10.1007/s11999-008-0209-4. Epub 2008 Apr 18. PMID 18421542
- [Background] Peel TN, Dowsey MM, Daffy JR, Stanley PA, Choong PF, Buising KL. Risk factors for prosthetic hip and knee infections according to arthroplasty site. J Hosp Infect. 2011 Oct;79(2):129-33. doi: 10.1016/j.jhin.2011.06.001. Epub 2011 Aug 6. PMID 21821313
- [Background] Rasouli MR, Restrepo C, Maltenfort MG, Purtill JJ, Parvizi J. Risk factors for surgical site infection following total joint arthroplasty. J Bone Joint Surg Am. 2014 Sep 17;96(18):e158. doi: 10.2106/JBJS.M.01363. PMID 25232088
- [Background] Karlakki S, Brem M, Giannini S, Khanduja V, Stannard J, Martin R. Negative pressure wound therapy for managementof the surgical incision in orthopaedic surgery: A review of evidence and mechanisms for an emerging indication. Bone Joint Res. 2013 Dec 18;2(12):276-84. doi: 10.1302/2046-3758.212.2000190. Print 2013. PMID 24352756
- [Background] Cooper HJ, Bas MA. Closed-Incision Negative-Pressure Therapy Versus Antimicrobial Dressings After Revision Hip and Knee Surgery: A Comparative Study. J Arthroplasty. 2016 May;31(5):1047-52. doi: 10.1016/j.arth.2015.11.010. Epub 2015 Nov 26. PMID 26712346
- [Background] Grauhan O, Navasardyan A, Hofmann M, Muller P, Stein J, Hetzer R. Prevention of poststernotomy wound infections in obese patients by negative pressure wound therapy. J Thorac Cardiovasc Surg. 2013 May;145(5):1387-92. doi: 10.1016/j.jtcvs.2012.09.040. Epub 2012 Oct 27. PMID 23111014

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevena: Subjects will receive PREVENA after surgery.
  Prevena: Closed Incision Negative Pressure Therapy (bandage over the incision sealed with negative pressure of a vacuum) to be placed on after surgery for 7 days.
  Prevena™, by KCI, is currently being used selectively in high-risk patients and a FDA-approved device.
- Aquacel: Subjects will receive AQUACEL Ag after surgery.
  Aquacel: Water resistant, silver-impregnated, antimicrobial hydrofiber dressing that is placed on after surgery for 7 days.
  AQUACEL® Ag, by Convatec, is currently the standard of care for postoperative wound dressing and a FDA-approved device.
Period: Overall Study
Arm/Group | Prevena | Aquacel
Started | 61 | 61
Completed | 60 | 60
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: 2 out of the 122 enrolled participants did not complete the study and therefore were not included in the data analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena | Aquacel | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 27 | 60
  >=65 years | 27 | 33 | 60
Age, Continuous [Mean (Full Range); unit: years] | 63.6 [32.8 to 85.9] | 64.4 [19 to 84.1] | 64 [19 to 85.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 21 | 23 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 2 | 5
  United States | 57 | 58 | 115

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Wound Complications
Description: Occurrence of wound complications (wound drainage, breakdown, necrosis, dehiscence, superficial or deep infection) requiring additional intervention. Intervention will be defined as any attempt of the surgeon to improve wound healing (in-office debridement, topical ointment, aspiration, antibiotic therapy, or return to the OR for the wound).
Time Frame: Up to 90 days
Population: 2 out of the 122 enrolled participants did not complete the study and therefore were not included in the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Aquacel
Number analyzed (Participants) | 60 | 60
Participants | 5 | 11

2. Secondary Outcome: Number of Patients With Superficial Surgical Site Infections
Description: Number of patients who met CDC criteria for superficial surgical site infection (SSI).
Time Frame: 90 days
Population: 2 out of the 122 enrolled participants did not complete the study and therefore were not included in the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Aquacel
Number analyzed (Participants) | 60 | 60
Participants | 2 | 9

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Prevena | Aquacel
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60
Other Adverse Events (participants affected / at risk) | 5/60 | 11/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena (N=60) | Aquacel (N=60)
Acute periprosthetic joint infection (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena (N=60) | Aquacel (N=60)
Surgical site complications (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (11) — Skin dehiscence to the subcutaneous level or prolonged drainage beyond five days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT03061903/Prot_SAP_000.pdf